CLINICAL TRIAL: NCT02500446
Title: Dolutegravir Impact on Residual Replication: Dolutegravir Intensification Study
Brief Title: Dolutegravir Impact on Residual Replication
Acronym: DIORR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: The Alfred (Other); ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Sharon Lewin, Director, Doherty Institute, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIORR_20150306
Record Dates: First submitted 2015-06-30; First posted 2015-07-16 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: HIV
MeSH Terms: interventions — dolutegravir

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Intensification (Active Comparator): Oral dolutegravir 50 mg once daily for 8 weeks added to their current ART regimen.
  Interventions: Drug: dolutegravir
- Placebo (Placebo Comparator): Oral placebo once daily for 8 weeks added to their current ART regimen.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: dolutegravir — Each film-coated tablet contains dolutegravir sodium equivalent to 50 mg dolutegravir.
  Other Names: Tivicay®
  Arms: Intensification
Other: Placebo — A film-coated tablet identical in appearance to the active drug tablet but not containing any dolutegravir or any other active ingredient
  Arms: Placebo

SUMMARY:
Several studies have suggested that despite suppressive combination antiretroviral therapy (ART) in people who are HIV-positive, in some individuals there may be on-going viral replication. Clarifying the extent of on-going viral replication on ART is important for the development of HIV-1 curative strategies and for reducing HIV-1 associated immune activation. The investigators hypothesize that treatment intensification with dolutegravir will inhibit residual virus replication in HIV-1 infected patients on ART. The primary objective of this study is to determine the effects of dolutegravir intensification on residual virus replication in circulating cluster of differentiation 4 (CD4+) T cells.

DETAILED DESCRIPTION:
ART effectively suppresses HIV-1 viremia but in most patients, virus rebounds within 2-3 weeks of stopping ART. ART is unable to cure HIV due to the persistence of virus as long-lived latently infected cells, residual virus replication and anatomical reservoirs. Understanding the contribution of residual virus replication to virus persistence on ART is important because first, no interventions aimed at eliminating latency will be effective in the presence of residual virus replication; second, residual virus replication may contribute to persisting immune activation which has been associated with all-cause mortality.

Numerous studies have demonstrated that intensifying a suppressive ART regimen with an additional antiretroviral drug does not alter the frequency of latently infected cells or low-level viremia. However, in studies that have intensified ART with the integrase inhibitor raltegravir, an increase in circularised HIV episomes containing 2 copies of the viral long terminal repeat (2-LTR) circles within 2 weeks of intensification, was observed in ~30% of study participants. 2-LTR circles have a short half- life, which may explain why an increase in 2-LTR circles was only observed in studies that measured 2-LTR circles within 2 weeks of raltegravir intensification. In these two randomized controlled trials, the level of 2-LTR circles increased transiently in patients randomized to intensification with raltegravir as compared with placebo and this effect was more pronounced in subjects receiving a protease inhibitor (PI)-containing ART regimen. Other studies have failed to demonstrate an increase in 2-LTR circles following raltegravir intensification but this is likely because sampling was delayed beyond 2 weeks.

One possible explanation for the additional effect observed with raltegravir intensification is the extensive penetration of this compound into gastrointestinal (GI) tissue where it reaches concentrations 39- to 650-fold higher than those in plasma.

To date, raltegravir is the only integrase inhibitor that has been investigated in ART intensification trials. Dolutegravir (DTG) is a recently licensed once-daily integrase inhibitor that is non-inferior to raltegravir and with a similar safety profile, however DTG levels in GI tissue is only 17% of that in plasma. DTG has not been investigated in intensification studies, so whether adding dolutegravir to a suppressive ART regimen is able to inhibit residual replication is currently unknown.

Thus, there are several unresolved issues related to residual viral replication in the presence of ART and the potential benefit of integrase inhibitors in this context: How frequent is this phenomenon and does it occur more frequently in patients receiving a PI-containing regimen? Given that raltegravir does seem to impact residual replication in approximate 30% of HIV infected patients on ART when assessed early after intensification, what is the effect of DTG in this setting? Finally, what are the dynamics of 2-LTR levels in blood in the early phases after intensification with an integrase inhibitor? To address those questions, the investigators have designed a randomized, controlled study to compare the impact of intensification with DTG or placebo in HIV-infected patients on suppressive ART. In this study, the investigators will closely define the effects of dolutegravir intensification on 2-LTR levels in circulating CD4+ T cells.

Study participants will be in the study for up to 133 days. The duration of participation is calculated from the initial screening visit to the last study visit (visit 9), with 9 visits in total.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Minimum age 18 years
* Receiving combination ART (at least 3 agents) for at least 3 years. Twenty of the 40 study participants will be on a PI-based ART regimen.
* HIV-1 plasma RNA <50 copies/mL for >3 years and <20 copies/mL at screening.
* Two CD4+ T cell counts >350 cells/μL in the 24 months prior to screening
* Able to give informed consent
* A female, may be eligible to enter and participate in the study if she:

  * Is of non-child-bearing potential OR
  * Is of child-bearing potential with a negative pregnancy test at both Screening and Day 1 and agrees to use one of the study protocol-specified methods of contraception to avoid pregnancy:

Exclusion Criteria:

* Known hypersensitivity to DTG or to any of the excipients
* Current use of dofetilide, pilsicainide or metformin
* Current use of etravirine except when etravirine is co-administered with atazanavir/ritonavir, lopinavir/ritonavir or darunavir/ritonavir
* Current or prior use of any integrase inhibitor
* Previous use of histone deacetylase inhibitors or other latency reversing agents
* Any significant acute medical illness requiring hospitalization within preceding 8 weeks
* Significant renal disease (eGFR <50 milliliters per min)
* Hepatitis C co-infection (Individuals with prior hepatitis C infection that is now cleared are eligible for enrolment)
* Subjects with severe hepatic impairment (Class C) as determined by Child-Pugh classification
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Receipt of immunomodulating agents (excluding immunization) or systemic chemotherapeutic agents within 28 days prior to study entry
* Patients who intend to modify their ART regimen within the study period
* Current or recent gastrointestinal disease or surgery that may impact the absorption of the investigational drug
* Active alcohol or substance use that in the opinion of the investigator will prevent adequate compliance with study procedures
* Currently pregnant, breastfeeding or unwilling to use barrier contraception
* Women of Child Bearing Potential (WOCBP) unwilling or unable to use an acceptable method of contraception to avoid pregnancy as specified in the inclusion criteria
* Unable or unwilling to adhere to protocol procedures
* The following laboratory values within 3 weeks before starting the investigational drug (lab tests may be repeated to obtain acceptable values before failure at screening is concluded)

  * Hepatic transaminases (AST or ALT) ≥3 x upper limit of normal (ULN)
  * Serum total bilirubin ≥1.5 x ULN
  * eGFR <50 mL/min
  * Haemoglobin <11.0 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2016-09-16 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Level of residual HIV replication in circulating CD4+ T cells | day 7 of treatment
  Change in the level of 2-LTR circles as measured by polymerase chain reaction (PCR) in the dolutegravir arm versus the placebo arm after 7 days of treatment

SECONDARY OUTCOMES:
Level of Human Leukocyte Antigen D-related (HLA-DR) | time points to day 84 (28 days after treatment)
  Change in level of Human Leukocyte Antigen D-related (HLA-DR), a marker of T cell activation from baseline within and across study arms.
Level of Programmed cell death-1 receptor (PD-1) | time points to day 84 (28 days after treatment)
  Change in level of Programmed cell death-1 receptor (PD-1), a marker of T cell activation from baseline within and across study arms.
Level of Cluster of Differentiation 38 (CD-38) | time points to day 84 (28 days after treatment)
  Change in level of Cluster of Differentiation 38 (CD-38), a marker of T cell activation, from baseline within and across study arms.
Level of residual HIV replication in circulating CD4+ T cells in a protease inhibitor -containing regimen | time points up to day 84 (28 days after treatment)
  Change in the level of 2-LTR circles as measured by polymerase chain reaction (PCR) in the dolutegravir arm versus the placebo arm in those participants on regimen which includes a protease inhibitor

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Lewin, Principal Investigator — Doherty Institute for Immunity and Infection
Locations (2):
- Australia (2):
  - Melbourne Sexual Health Centre, Carlton, Victoria
  - Alfred Hospital, Prahran, Victoria

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data

REFERENCES:
- [Derived] Rasmussen TA, McMahon JH, Chang JJ, Audsley J, Rhodes A, Tennakoon S, Dantanarayana A, Spelman T, Schmidt T, Kent SJ, Morcilla V, Palmer S, Elliott JH, Lewin SR. The effect of antiretroviral intensification with dolutegravir on residual virus replication in HIV-infected individuals: a randomised, placebo-controlled, double-blind trial. Lancet HIV. 2018 May;5(5):e221-e230. doi: 10.1016/S2352-3018(18)30040-7. Epub 2018 Apr 8. PMID 29643011